CLINICAL TRIAL: NCT00411320
Title: Determinants of Corticosteroid Insensitivity in Smokers With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: Chief Scientist Office of the Scottish Government (Other Government)
Responsible Party: Dr Caroline Watson, R&D Manager, NHS Greater Glasgow and Clyde (North Glasgow University Hospitals Division)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AR002
Record Dates: First submitted 2006-12-12; First posted 2006-12-14 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2008-09

CONDITIONS: Asthma; Smoking; Steroid Resistance; Corticosteroid Insensitivity
Keywords: Asthma; Smoking; Steroid Resistance; Corticosteroid insensitivity
MeSH Terms: conditions — Asthma; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group 1 (Active Comparator): Smokers with asthma
  Interventions: Drug: oral steroid-dexamethasone
- Group 2 (Active Comparator): Ex-smokers with asthma
  Interventions: Drug: oral steroid-dexamethasone
- Group 3 (Active Comparator): Non-smokers with asthma
  Interventions: Drug: oral steroid-dexamethasone
- Group 4 (No Intervention): Non smokers without asthma
- Group 5 (No Intervention): Smokers without asthma or COPD

INTERVENTIONS:
Drug: oral steroid-dexamethasone — 2 week steroid trial
  Arms: Group 1; Group 2; Group 3

SUMMARY:
Smokers with asthma display a relative insensitivity to inhaled and oral corticosteroids. The causes of this phenomenon are currently unknown. The investigators will perform a number of blood & breathing tests to try to discover the cause/s behind this phenomenon with the aim of producing leads for further investigation and possible new treatments for smokers with asthma.

DETAILED DESCRIPTION:
Smokers with asthma display a relative insensitivity to inhaled and oral corticosteroids. The causes of this phenomenon are currently unknown. However research into steroid resistance in severe asthma and the smoking related condition chronic obstructive pulmonary disease (COPD) points to a number of possible causes. We will characterise a group of smokers with asthma and perform a number of investigations and compare the results to ex-smokers and never smokers with asthma with the aim of establishing which previously published steroid resistance phenomena are related to the steroid resistance displayed by smokers with asthma. Results produced from this trial will provide hypothesis generating information leading to future pharmaceutical trials.

ELIGIBILITY:
Inclusion Criteria:

* Asthma (defined by either reversibility to bronchodilator or methacholine testing)
* Asthma duration of 6 months or greater
* Stable asthma
* Age 18-60
* Treatment with inhaled corticosteroids
* Smoking history consistent with group

  * smokers with asthma: > or = 5 pack years and currently smoking more than 5 cigarettes per day
  * ex-smokers: smoking ceased > or = two years prior to recruitment, minimum 5 pack year history
  * non-smokers: no smoking history

Exclusion Criteria:

* Presence of medical condition likely to be exacerbated by treatment with oral corticosteroids
* Treatment with > 2000 mcg beclomethasone (or equivalent) per day
* Subject requires oral corticosteroids to maintain asthma control
* Subject requires oral theophylline to maintain asthma control
* Recent treatment with oral corticosteroids
* Pregnancy or subject planning to become pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2007-01; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
bronchodilator response to oral corticosteroid trial in smokers with asthma vs non smokers and ex-smokers with asthma | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark Spears, MRCP, Principal Investigator — University of Glasgow; Neil C Thomson, FRCP, Principal Investigator — University of Glasgow; Rekha Chaudhuri, MD, Principal Investigator — University of Glasgow
Locations (1):
- Asthma Research Unit, Glasgow University, Glasgow, Scotland, United Kingdom

REFERENCES:
- [Derived] Spears M, McSharry C, Donnelly I, Jolly L, Brannigan M, Thomson J, Lafferty J, Chaudhuri R, Shepherd M, Cameron E, Thomson NC. Peripheral blood dendritic cell subtypes are significantly elevated in subjects with asthma. Clin Exp Allergy. 2011 May;41(5):665-72. doi: 10.1111/j.1365-2222.2010.03692.x. Epub 2011 Feb 21. PMID 21338429
- See also: unit website — http://www.gla.ac.uk/departments/immunology/respiratorymedicine/